CLINICAL TRIAL: NCT06307145
Title: Efficacy and Safety of Hip Replacement Surgery Using Korean National Registry
Brief Title: Korea Hip Replacement Surgery Registry
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Juhee Cho, Professor, Samsung Medical Center
Other Study IDs: K-NHIS-HIP
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Hip Replacement Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This cohort study obtained data from the Korean National Health Insurance Service (K-NHIS) database. For the hip replacement registry, we included all adult patients older than 19 who received total or hemiarthroplasty surgery between January 1, 2003, and December 31, 2019. Using this registry, we compared efficacy and safety by type of head or liner.

DETAILED DESCRIPTION:
This cohort study obtained data from the Korean National Health Insurance Service (K-NHIS) database. For the hip replacement registry, we included all adult patients older than 19 who received total or hemiarthroplasty surgery between January 1, 2003, and December 31, 2019. Using this registry, we compared efficacy and safety by type of head or liner. The safety issues included the incidence of cancer, orthoperiodic outcome (dislocation, mechanical Cx, periprosthetic join infection, periprosthetic fracture), revision, embolism or thrombosis, cardiac outcome, and death

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 19 or older who received hip replacement surgery

Exclusion Criteria:

* Insufficient information
* history of any revision

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient aged 19 or older who received hip replacement surgery
Sampling Method: Non-Probability Sample
Enrollment: 124556 (Actual)
Dates: Start 2003-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Cancer | the occurrence of cancer, death, or December 31st, 2019 (end of the study), whichever came first.
  Incidence of cancer

CONTACTS AND LOCATIONS:
Overall Officials: Juhee Cho, Principal Investigator — Samsung Medical Center

IPD SHARING:
Plan to Share IPD: No
Access to the dataset is limited to researchers who have been approved by the NHIS.